CLINICAL TRIAL: NCT03205904
Title: Nutritional Intervention and Glycemic Improvement in Patients With Pre-diabetic Cystic Fibrosis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 160206
Record Dates: First submitted 2017-06-15; First posted 2017-07-02 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Cystic Fibrosis-related Diabetes; Cystic Fibrosis
Keywords: cystic fibrosis related diabetes
MeSH Terms: conditions — Cystic Fibrosis | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Group that will be receive the diet
  Interventions: Dietary Supplement: Diet
- control (No Intervention): Group that will not receive the diet

INTERVENTIONS:
Dietary Supplement: Diet — Nutrition booklet with guidelines on types of fats and glycemic index
  Arms: Intervention group

SUMMARY:
Cystic fibrosis (CF) is a genetic disease with an autosomal recessive, chronic and progressive character about 10 to 25% of patients develop CF-related diabetes (DRFC). Until now, there is no evidence to support the use of low glycemic index diet to improve glycemic response in pre-diabetic and CF patients. The objective of this study is to evaluate the glycemic improvement after nutritional orientation in patients with cystic fibrosis.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is a genetic disease with an autosomal recessive, chronic and progressive character. About 10 to 25% of patients develop CF-related diabetes (DRFC), whose pathogenesis is associated with pancreatic fibrosis and destruction. Until now, there is no evidence to support the use of low glycemic index diet to improve glycemic response in pre-diabetic and CF patients. The objective of this study is to evaluate the glycemic improvement after nutritional orientation in patients with cystic fibrosis in the pre-diabetic phase. Methods: Randomized clinical trial in patients with CF aged over 10 years without hospitalization in the last 4 weeks. Anthropometric measurements, blood pressure, 24 hour recall and food frequency questionnaire will be evaluated. Oral glucose tolerance and glycated hemoglobin test will be dosed at baseline and during 12 weeks of follow-up. The intervention group will receive a nutritional guidance at the beginning of the research.

ELIGIBILITY:
Inclusion Criteria:

* tolerance glucose test values between 100 and 125mg / dl and or glucose 2h after 75g of glucose between 140 and 199 mg / dl
* Stable pulmonary disease in the last four weeks

Exclusion Criteria:

* Without hospitalization in the last 3 months

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
glycemic improvement after nutritional orientation in patients with cystic fibrosis in the pre-diabetic phase | 3 months
  To evaluate the improvement of glucose levels after the diet intervention. After 12 weeks of intervention will be performed oral glucose tolerance test

SECONDARY OUTCOMES:
Evaluate the levels of HbA1c before and after the intervention | 3 months
  Evaluate the levels of HbA1c before and after the intervention
Evaluate the response of forced expiratory volume and forced vital capacity before and after the intervention | 3 months
  Evaluate the response of FEV 1 (forced expiratory volume) before and after the intervention
To evaluate anthropometric data of the patients before and after the intervention. | 3 months
  Improvement of nutritional status Using weight (kg) and height (cm) and BMI.

CONTACTS AND LOCATIONS:
Overall Officials: Ticiana C Rodrigues, Doctor, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Ticiana da Costa Rodrigues, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No